CLINICAL TRIAL: NCT00388882
Title: A Randomized, Double-blind, Double-dummy, Parallel Group Trial Comparing 12 Weeks Treatment With Tiotropium Inhalation Capsules 18 mcg Via the HandiHaler® Once Daily to Combivent® Inhalation Aerosol CFC MDI 2 Actuations q.i.d. in COPD Patients Currently Prescribed Combivent® Inhalation Aerosol CFC MDI
Brief Title: Trial Comparing Treatment With Tiotropium Inhalation Capsules to Combivent® Inhalation Aerosol in COPD Patients.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 205.346; EudraCT 2006-000822-30
Record Dates: First submitted 2006-10-16; First posted 2006-10-17 (Estimated); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; Ipratropium; Albuterol

INTERVENTIONS:
Drug: tiotropium
Drug: ipratropium bromide / albuterol

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of 12 weeks treatment with tiotro pium HandiHaler® 18 mcg daily compared to Combivent® MDI CFC Inhalation Aerosol 2 actuations qid in COPD patients currently prescribed Combivent® MDI.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD
* Age: >= 40 years
* Current or ex-smoker with a >= 10 pack-year smoking history
* Use of Combivent® MDI for >= 1 month prior to Visit 1 Spirometric criteria (determined at study visits):
* Post-bronchodilator FEV1 <= 70% (Visit 1)
* Pre-bronchodilator FEV1 <= 65% of predicted and FEV1/FVC <= 70% (Visit 2)

Exclusion Criteria:

* Clinical history of asthma
* History of thoracotomy with pulmonary resection
* History of CF, alpha 1 antitrypsin deficiency or interstitial lung disease
* Daytime use of oxygen therapy for > 1 hour per day or if unable to abstain from using oxygen during PFTs
* Any respiratory tract infection or COPD exacerbation in 6 weeks prior to Visit 1
* Recent history 6 months or less of MI
* Unstable or life-threatening cardiac arrhythmias
* Hospitalization for CHF during past year
* Malignancy for which patient is receiving chemo or radiation therapy
* Pregnant or nursing women
* Known hypersensitivity to ipratropium or carrier substances, including related food products such as soybean, peanuts, or lactose
* Use of SPIRIVA® 3 months prior to Visit 1
* Symptomatic of prostatic hypertrophy or bladder neck obstruction
* Known narrow- angle glaucoma
* Participating in a pulmonary rehab program within 4 weeks of Visit 1

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2006-10-04 (Actual); Primary Completion 2007-10-08 (Actual)

PRIMARY OUTCOMES:
Trough FEV1 | after 12 weeks of treatment
FEV1 AUC0-6 hours | after 12 weeks of treatment

SECONDARY OUTCOMES:
Peak FEV1 | 12 weeks
Peak FEV1 | after first dose and 6 week
FEV1 AUC0-6 hours | after first dose and 6 weeks
Trough FEV1 | at 6 weeks
Peak FVC at all clinic visits | 12 weeks
AUC0-6 hours FVC at all clinic visits | 12 weeks
Trough FVC | at 6 and 12 weeks
Individual FEV1 measurements | 12 weeks
Individual FVC measurements | 12 weeks
Use of Albuterol (scheduled and rescue) | 12 weeks
Patient Global Evaluation | 12 weeks
Physician Global Evaluation | 12 weeks
PEFR (Peak expiratory flow rate) measured by the patient at home twice daily | 12 weeks
Occurrence of adverse events | 12 weeks
Vital Signs | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (40):
- United States (10):
  - 205.346.107 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 205.346.104 Boehringer Ingelheim Investigational Site, Lakewood, California
  - 205.346.108 Boehringer Ingelheim Investigational Site, Sepulveda, California
  - 205.346.101 Boehringer Ingelheim Investigational Site, Torrance, California
  - 205.346.106 Boehringer Ingelheim Investigational Site, Wheat Ridge, Colorado
  - 205.346.102 Boehringer Ingelheim Investigational Site, Coeur d'Alene, Idaho
  - 205.346.109 Boehringer Ingelheim Investigational Site, Shreveport, Louisiana
  - 205.346.110 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 205.346.105 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 205.346.103 Boehringer Ingelheim Investigational Site, Spartanburg, South Carolina
- Argentina (8):
  - 205.346.510, Bs As
  - 205.346.502, Buenos Aires
  - 205.346.503, Buenos Aires
  - 205.346.508, Buenos Airess
  - 205.346.505, Mendoza
  - 205.346.509, Rosario, Santa Fe
  - 205.346.511, Rosario, Santa Fé
  - 205.346.504 Instituto de Patologías Respiratorias, San Miguel de Tucumán
- Lithuania (9):
  - 205.346.401 Boehringer Ingelheim Investigational Site, Alytus
  - 205.346.404 Boehringer Ingelheim Investigational Site, Kaunas
  - 205.346.405 Boehringer Ingelheim Investigational Site, Kaunas
  - 205.346.411 Boehringer Ingelheim Investigational Site, Klaipėda
  - 205.346.409 Boehringer Ingelheim Investigational Site, Šiauliai
  - 205.346.408 Boehringer Ingelheim Investigational Site, Utena
  - 205.346.402 Boehringer Ingelheim Investigational Site, Vilnius
  - 205.346.406 Boehringer Ingelheim Investigational Site, Vilnius
  - 205.346.407 Boehringer Ingelheim Investigational Site, Vilnius
- Slovakia (6):
  - 205.346.302 Boehringer Ingelheim Investigational Site, Bratislava
  - 205.346.305 Boehringer Ingelheim Investigational Site, Bratislava
  - 205.346.301 Boehringer Ingelheim Investigational Site, Košice
  - 205.346.303 Boehringer Ingelheim Investigational Site, Levica
  - 205.346.304 Boehringer Ingelheim Investigational Site, Lučenec
  - 205.346.306 Boehringer Ingelheim Investigational Site, Štúrovo
- United Kingdom (7):
  - 205.346.204 Boehringer Ingelheim Investigational Site, Aylesbury
  - 205.346.203 Boehringer Ingelheim Investigational Site, Greenisland
  - 205.346.201 Boehringer Ingelheim Investigational Site, Nottingham
  - 205.346.207 Boehringer Ingelheim Investigational Site, Soham
  - 205.346.209 Boehringer Ingelheim Investigational Site, Swansea
  - 205.346.206 Boehringer Ingelheim Investigational Site, Westbury on Trym
  - 205.346.205 Boehringer Ingelheim Investigational Site, Windsor

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/19737620